CLINICAL TRIAL: NCT05947851
Title: A Phase 3, Open-label, Randomized Study to Compare the Efficacy and Safety of Nemtabrutinib (MK-1026) Plus Venetoclax Versus Venetoclax Plus Rituximab in Participants With Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma Following at Least 1 Prior Therapy (BELLWAVE-010)
Brief Title: A Study of Nemtabrutinib Plus Venetoclax vs Venetoclax + Rituximab (VR) in Second-line (2L) + Relapsed/Refractory (R/R) Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) (MK-1026-010/BELLWAVE-010).
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1026-010; MK-1026-010 (Other: MSD); BELLWAVE-010 (Other: MSD); 2022-501560-17-00 (Registry Identifier: EU CT); U1111-1281-1520 (Registry Identifier: UTN)
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Chronic Lymphocytic; Small-Cell Lymphoma; Lymphoma, Small Lymphocytic; CLL; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ARQ531; venetoclax; Rituximab

STUDY DESIGN:
Intervention Model Description: In Part 1, Dose Confirmation will be determined by modified toxicity probability interval (mTPI) design, where participants will be assigned to two treatment groups, Nemtabrutinib + Venetoclax in parallel with Nemtabrutinib + Venetoclax. Part 2 will be an Efficacy Expansion where all participants will be randomized 1:1 to Nemtabrutinib Part 1 Dose Selection plus Venetoclax or Venetoclax plus Rituximab (VR) (or Rituximab biosimilar) for the duration of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nemtabrutinib + Venetoclax (Experimental): Participants will receive nemtrabrutinib oral tablets at specified doses daily starting at Cycle 1 Day 1 (C1D1) and venetoclax oral tablets at doses of 20 mg up to 400 mg daily starting at Cycle 2 Day 1 (C2D1) up to 2 years post C2D1 or until progressive disease (PD) or discontinuation. A cycle = 4 weeks.
  Interventions: Drug: Nemtabrutinib; Drug: Venetoclax
- Venetoclax + Rituximab (Active Comparator): Participants will receive venetoclax oral tablets at doses from 20 mg up to 400 mg daily starting at C1D1 on 4-week cycles up to 2 years and rituximab or biosimilar at 375 mg/m^2 up to 500 mg/m2 intravenous infusion once per 28-day cycle starting at C2D1, for 6 total cycles. Treatment will continue until progressive disease (PD) or discontinuation.
  Interventions: Drug: Venetoclax; Biological: Rituximab

INTERVENTIONS:
Drug: Nemtabrutinib — 5, 20, 45, and 65 mg tablets
  Other Names: ARQ 531; MK-1026
  Arms: Nemtabrutinib + Venetoclax
Drug: Venetoclax — 10, 50, and 100 mg tablets
  Other Names: ABT-199; GDC-0199
Biological: Rituximab — 100 mg/10 mL, 500 mg/50 mL (10 mg/mL) IV Infusion
  Arms: Venetoclax + Rituximab

SUMMARY:
The purpose of this study is to assess the safety and tolerability and to confirm the dose of nemtabrutinib in combination with venetoclax in participants with R/R CLL/SLL. The primary study hypotheses are that the combination of nemtabrutinib plus venetoclax is superior to VR with respect to progression-free survival (PFS) per 2018 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria as assessed by blinded independent central review (BICR).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) and active disease clearly documented to initiate therapy
* Deletion (Del) (17p) status, tumor protein 53 (TP53) mutation status, and immunoglobulin heavy chain gene (IGHV) mutation status results required before randomization for Part 2 participants only
* Relapsed or refractory to at least 1 prior available therapy
* Have at least 1 marker of disease burden
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 within 7 days before randomization
* Has a life expectancy of at least 3 months
* Has the ability to swallow and retain oral medication
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV deoxyribonucleic acid (DNA) viral load before randomization
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV ribonucleic acid (RNA) viral load is undetectable at screening
* Participants with human immunodeficiency virus (HIV) who meet ALL eligibility criteria
* Participants with adequate organ function with specimens collected within 7 days before the start of study intervention
* If capable of producing sperm, participant agrees to eliminate Nemtabrutinib: 12 days, Venetoclax: 1 month (30 days), Rituximab (rituximab biosimilar): not applicable; abstains from penile-vaginal intercourse as their preferred and usual lifestyle; OR uses prescribed contraception
* Participant assigned female sex at birth are eligible to participate if not pregnant or breastfeeding and are not a person of childbearing potential (POCBP) OR is a POCBP and uses a contraceptive method that is highly effective, has a negative highly sensitive pregnancy test, and abstains from breastfeeding

Exclusion Criteria:

* Has an active hepatitis B virus/ hepatitis C virus (HBV/HCV) infection
* Has gastrointestinal (GI) dysfunction that may affect drug absorption
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years
* Has diagnosis of Richter Transformation or active central nervous system (CNS) involvement by CLL/SLL
* Has an active infection requiring systemic therapy, such as intravenous (IV) antibiotics, during screening
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease and/or acquired immune deficiency syndrome (AIDS)-defining opportunistic infection in the past 12 months before screening
* Clinically significant cardiovascular disease
* Has a known allergy/sensitivity to nemtabrutinib or contraindication to venetoclax/rituximab (or rituximab biosimilar), or any of the excipients
* Has history of severe bleeding disorders (eg, hemophilia)
* Has received prior systemic anticancer therapy within 5 half-lives or 4 weeks (if prior therapy was a monoclonal antibody) before randomization
* Has received prior B-cell lymphoma 2 inhibitor(s) (BCL2i) within ≤ 12 months before randomization or has received prior radiotherapy within 2 weeks of start of study intervention, or radiation related toxicities, requiring corticosteroids
* Is currently being treated with p-glycoprotein (P-gp) substrates with a narrow therapeutic index, cytochrome P450 3A (CYP3A) strong or moderate inducers or CYP3A strong inhibitors.
* Has received a live or live attenuated vaccine within 30 days before the first dose of study intervention
* Has received an investigational agent or has used an investigational device within 4 weeks before study intervention administration
* Has a known psychiatric or substance use disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Participants who have not adequately recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 735 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2032-06-01 (Estimated); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants Experiencing Dose-Limiting Toxicities (DLTs) | Up to approximately 12 Weeks
  DLT evaluation period is defined as 8 weeks after the first dose of the combination treatment of nemtabrutinib plus venetoclax Cycle 2 Day 1 in Part 1 + 4 weeks follow up. Each cycle is 4 weeks. DLTs are: Grade ≥3 nonhematologic toxicity (except Grade 3 nausea, vomiting, diarrhea, rash, fatigue, and uncontrolled hypertension which will not be considered a DLT unless lasting ≥72 hours despite optimal supportive care); Grade 4 hematologic toxicity lasting >7 days (except Grade 3 lymphocytosis, Grade 4 platelet count decreased of any duration, or Grade 3 platelet count decreased if associated with bleeding); any Grade 3 or Grade 4 nonhematologic laboratory abnormality if values result in drug-induced liver injury, or medical intervention is required, or the abnormality leads to hospitalization, or the abnormality persists for >1 week (with exceptions); missing >25% of nemtabrutinib or venetoclax doses as a result of drug-related adverse events during the first 2 cycles; Grade 5 toxicity.
Part 1: Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 28 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants experiencing AEs will be reported for Part 1.
Part 1: Number of Participants Discontinuing Study Treatment Due to AEs | Up to approximately 25 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants discontinuing study treatment due to AEs will be reported for Part 1.
Part 2: PFS per the 2018 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Criteria as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 71 months
  PFS is defined as the time from randomization to the first documented disease progression per iwCLL criteria 2018 as accessed by BICR, or death due to any cause, whichever occurs first. PFS will be presented.

SECONDARY OUTCOMES:
Part 2: Undetectable Minimal Residual Disease (MRD) Rate in Bone Marrow as Assessed by Central Laboratory | Up to approximately 46 months
  Undetectable MRD, defined as <1 leukemic cell per 10,000 cells (MRD <10-4) in bone marrow. The MRD rate will be presented.
Part 2: Overall Survival (OS) | Up to approximately 108 months
  OS, defined as the time from randomization to death due to any cause. OS will be presented.
Part 2: Objective Response Rate (ORR) per iwCLL Criteria 2018 as Assessed by BICR | Up to approximately 71 months
  OR, defined as complete response/remission (CR), complete response with incomplete count recovery (CRi), nodular partial remission (nPR), or partial remission (PR). CR is defined as meeting the following criteria: no lymph nodes >1.5 cm, spleen size <13 cm, liver normal; no constitutional symptoms, normal lymphocyte count, platelets ≥100 x 10^9/L; hemoglobin ≥11 g/dL; and normocellular marrow (no CLL cells or B lymphoid nodules). CRi is defined as meeting CR criteria but with hypocellular bone marrow. nPR is defined as having features of CR but with lymphoid nodules in the marrow. PR is defined as ≥50% decrease in ≥2 of the following: lymph nodes, liver and/or spleen size, lymphocytes PLUS ≥1 of the following met: platelets ≥100 x 10^9/L or ≥50% increase from screening, hemoglobin >11 g/dL or ≥50% increase from screening, CLL cells or B lymphoid nodules in marrow. ORR will be presented.
Part 2: Duration of Response (DOR) per iwCLL Criteria 2018 as Assessed by BICR | Up to approximately 108 months
  DOR, defined as the time from the first documented evidence of CR, CRi, nPR, or PR that led to response until disease progression or death due to any cause, whichever occurs first. CR is defined as meeting the following criteria: no lymph nodes >1.5 cm, spleen size <13 cm, liver normal; no constitutional symptoms, normal lymphocyte count, platelets ≥100 x 10^9/L; hemoglobin ≥11 g/dL; and normocellular marrow (no CLL cells or B lymphoid nodules). CRi is defined as meeting CR criteria but with hypocellular bone marrow. nPR is defined as having features of CR but with lymphoid nodules in the marrow. PR is defined as ≥50% decrease in ≥2 of the following: lymph nodes, liver and/or spleen size, lymphocytes PLUS ≥1 of the following met: platelets ≥100 x 10^9/L or ≥50% increase from screening, hemoglobin >11 g/dL or ≥50% increase from screening, CLL cells or B lymphoid nodules in marrow. DOR will be presented.
Part 2: Number of Participants Experiencing AEs | Up to approximately 28 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants experiencing AEs will be reported for Part 2.
Part 2: Number of Participants Discontinuing Study Treatment Due to AEs | Up to approximately 25 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants discontinuing study treatment due to AEs will be reported for Part 2.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (52):
- United States (6):
  - Highlands Oncology Group ( Site 5405), Springdale, Arkansas
  - MemorialCare Health System - Long Beach Medical Center ( Site 5421), Long Beach, California
  - Memorial Hospital West ( Site 5410), Pembroke Pines, Florida
  - Oregon Health and Science University ( Site 5425), Portland, Oregon
  - Medical Oncology Associates, PS ( Site 5406), Spokane, Washington
  - University of Wisconsin Hospital and Clinics-Carbone Cancer Center ( Site 5423), Madison, Wisconsin
- Argentina (5):
  - Instituto Alexander Fleming ( Site 1005), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 1007), Mar del Plata, Buenos Aires
  - Sanatorio Parque ( Site 1003), Rosario, Santa Fe Province
  - Centro Medico Fleischer ( Site 1006), Buenos Aires
  - Hospital Aleman-oncohematologic diseases ( Site 1001), Buenos Aires
- Australia (2):
  - Royal Adelaide Hospital ( Site 1104), Adelaide, South Australia
  - Western Health-Sunshine & Footscray Hospitals-Cancer Services-Cancer Research ( Site 1103), Melbourne, Victoria
- Belgium (2):
  - UZ Leuven-Hematology ( Site 1200), Leuven, Vlaams-Brabant
  - ZAS Cadix ( Site 1203), Antwerp
- ICESP - INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO-Pesquisa Clinica ( Site 1308), São Paulo, Brazil
- The Moncton Hospital ( Site 1414), Moncton, New Brunswick, Canada
- Chile (5):
  - IC La Serena Research ( Site 1506), La Serena, Coquimbo Region
  - Centro de Estudios Clínicos SAGA-CECSAGA ( Site 1509), Santiago, Region M. de Santiago
  - FALP-UIDO ( Site 1500), Santiago, Region M. de Santiago
  - Clínica Inmunocel ( Site 1511), Santiago, Region M. de Santiago
  - Biocenter ( Site 1507), Concepción, Región del Biobío
- Fundación Valle del Lili ( Site 1703), Cali, Valle del Cauca Department, Colombia
- France (3):
  - Hopital Claude Huriez - CHU de Lille ( Site 2107), Lille, Nord
  - Centre Hospitalier Universitaire Estaing ( Site 2105), Clermont-Ferrand, Puy-de-Dome
  - CHD Vendee ( Site 2100), La Roche-sur-Yon, Vendee
- Germany (2):
  - Klinikum Mutterhaus der Borromäerinnen-Innere Medizin I ( Site 2203), Trier, Rhineland-Palatinate
  - Universitätsklinikum Leipzig-Medical Department I - Hematology and Celltherapy ( Site 2201), Leipzig, Saxony
- Israel (4):
  - Rambam Health Care Campus ( Site 2801), Haifa
  - Hadassah Medical Center-Hemato-Oncology ( Site 2812), Jerusalem
  - Sheba Medical Center-Hemato Oncology ( Site 2809), Ramat Gan
  - Sourasky Medical Center ( Site 2811), Tel Aviv
- Italy (3):
  - Azienda Ospedaliero-Universitaria SS. Antonio e Biagio e Cesare Arrigo ( Site 2906), Alessandria, Ancona
  - Ospedale San Raffaele-Programma di Ricerca Strategica sulla LLC ( Site 2902), Milan
  - Arcispedale Santa Maria Nuova-Hematology ( Site 2900), Reggio Emilia
- Mexico (3):
  - Centro de Infusion Superare ( Site 3314), Mexico City, Mexico City
  - Health Pharma Professional Research S.A. de C.V: ( Site 3301), Mexico City, Mexico City
  - Centro de Investigacion Clinica Chapultepec ( Site 3309), Morelia, Michoacán
- Auxilio Mutuo Cancer Center ( Site 3900), San Juan, Puerto Rico
- South Africa (3):
  - Alberts Cellular Therapy. ( Site 4401), Pretoria, Gauteng
  - Groote Schuur Hospital ( Site 4400), Cape Town, Western Cape
  - Haemalife ( Site 4407), Kuilsriver, Western Cape
- Spain (3):
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals-Haematology Department ( Site 4601), L'Hospitalet Del Llobregat, Barcelona
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID ( Site 4602), Pozuelo de Alarcón, Madrid
  - HOSPITAL CLINICO DE VALENCIA-HEMATOLOGY ( Site 4603), Valencia, Valenciana, Comunitat
- Turkey (Türkiye) (5):
  - Ege Universitesi Hastanesi ( Site 4902), Bornova, İzmir
  - Namik Kemal University Medical Faculty-Hematology ( Site 4912), Tekirdağ, Tekirdas
  - Ankara Universitesi Tip Fakultesi Hastanesi-hematology ( Site 4913), Ankara
  - Mega Medipol-Hematology ( Site 4904), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi ( Site 4906), Istanbul
- United Kingdom (2):
  - City Hospital, Nottingham University Hospitals-Hematology ( Site 5002), Nottingham, England
  - University College London Hospital-Cancer Clinical Trials Unit ( Site 5001), London-Camden, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26318&tenant=MT_MSD_9011